CLINICAL TRIAL: NCT06986096
Title: Lifestyle for the BRAin Health - Nutrition and Exercise Training Intervention, LIBRA-NET
Brief Title: Lifestyle for the BRAin Health - Nutrition and Exercise Training Intervention
Acronym: LIBRA-NET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Slovak Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Barbara Ukropcová, MD, PhD, Professor, Slovak Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 101087124
Record Dates: First submitted 2024-07-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Aging; Alzheimer Disease; Life Style, Healthy; Exercise; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Motor Activity; Cognitive Dysfunction | interventions — Nutrition Assessment; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: ID codes will be provided for the outcomes assessor, without group-specific characterization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic-strength training and nutritional counseling (Experimental): Elderly volunteers participating in aerobic-strength training and nutritional counseling.
  Interventions: Behavioral: Aerobic-strength training and nutritional counseling
- Cognitive training and stretching. (Experimental): Elderly volunteers participating in cognitive training combined with stretching training.
  Interventions: Behavioral: Cognitive training and stretching.

INTERVENTIONS:
Behavioral: Aerobic-strength training and nutritional counseling — The intervention consists of a structured program that includes aerobic-strength training (1h training, 3 times per week) conducted by professional trainers combined with nutritional counseling.
  Arms: Aerobic-strength training and nutritional counseling
Behavioral: Cognitive training and stretching. — The intervention consists of a structured program that includes cognitive training combined with stretching training (90mins training, 2x per week).
  Arms: Cognitive training and stretching.

SUMMARY:
Due to the increasing incidence of dementia and the lack of causal treatment, non-pharmacological interventions represent an attractive and effective therapeutic strategy of neurodegenerative diseases, such as Alzheimer's disease.

The aim of the study is to assess the impact of a supervised 9-month intervention with aerobic-strength training and nutritional counseling compared to cognitive training and stretching on the brain, cognitive and motor functions, metabolism, physical fitnes and plasma markers of neurodegenertion in older adults at increased risk of developing Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Signed informed consent
* Presence of subjective or mild cognitive impairment (SCI/aMCI)
* Elevated levels of selected biomarkers confirming the presence of a pathological process characteristic of Alzheimer's disease
* Absence of any psychological, sociological, or geographical factors that could jeopardize participation in the project.

Exclusion Criteria:

* Presence of severe cardiovascular, liver, or kidney diseases; advanced or poorly controlled diabetes mellitus (HbA1c >7%), treated with insulin or incretin analogs; cancer or any other severe disease as assessed by the responsible physician. A history of cancer treated with chemotherapy or radiotherapy if within less than 5 years post-treatment.
* Lack of cooperation, inflexible schedule, or problematic transportation.
* Insufficient functional capacity or presence of comorbidities that prevent participation in the training program (assessment by an internist, cardiologist, neurologist, orthopedic specialist, or other relevant specialists).
* Presence of a pacemaker or any metal implants (contraindication for MRI examination), or allergy to local anesthetics (contraindication for muscle biopsy).
* Smoking, alcohol dependence, or addiction to other narcotic substances.
* Stroke or myocardial infarction within the last year.
* Long-term treatment for psychiatric disorders - a depressive syndrome is not an exclusion criterion if it is compensated by therapy.
* Other diseases of the musculoskeletal or nervous system that potentially interfere with the ability to exercise or cognition - such as severe arthritis, Parkinson's disease, significant essential tremor, epilepsy, etc.
* Concurrent participation in another clinical study.
* Therapy with cholinesterase inhibitors unless the patient is on a stable dose.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Impact on Cognitive Functions | Measurements at the baseline and after 9-month intervention.
  Overall composite score of neuropsychological testing batery (higher score better outcome)
Effect of Interventions on Neurodegeneration Markers | Measurements at the baseline and after 9-month intervention
  Concentration of plasma neurodegeneration marker pTau 217 (in a subpopulation of patients).

SECONDARY OUTCOMES:
Computerized Cognitive Tests | Measurements at the baseline and after 9-month intervention.
  Computerised cognitive testing CogState (learning/working memory score, higher score - better outcome)
Well-being | Measurements at the baseline and after 9-month intervention.
  The World Health Organization Quality of Life questionaire (WHOQOL-BREF), 31 items, highre score better QoL.
Glucose metabolism | Measurements at the baseline and after 9-month intervention.
  oral glucose tolerance test will be perfromed to detect level of glucose intolerance (impaired glucose tolerance)
MRI of the Brain | Measurements at the baseline and after 9-month intervention.
  Imaging studies to assess structural adaptation of the brain (hippocampal volume).
Adherence | Adherence will be recorded during the 9-month intervention period.
  Evaluation of participant adherence to the intervention protocol.
Olfactory Function | Measurements at baseline and after 9-month intervention.
  Olfactory function screening test (The Sniffin' Sticks test kit).
Microbiome Composition | Measurements at baseline and after 9-month intervention.
  Determination of feacal microbiome composition (16S sequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Ukropcova, Prof., Principal Investigator — Biomedical Research Center Slovak Academy of Science
Locations (1):
- Biomedical Research Center Slovak Academy of Sciences, Bratislava, Bratislava Region, Slovakia

IPD SHARING:
Plan to Share IPD: No